CLINICAL TRIAL: NCT03420534
Title: Human Bioequivalence Test (Fasting & Postprandial) of Iloperidone Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDY2017002
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Bioequivalence
MeSH Terms: interventions — iloperidone; Angptl4 protein, mouse; Postprandial Period

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- iloperidone in fasting (Experimental): iloperidone 1mg by mouth once for 6 days in the first cycle or the second cycle
  Interventions: Drug: Iloperidone 1 MG; Dietary Supplement: fasting
- placebo tablets in fasting (Active Comparator): placebo mimic iloperidone 1mg by mouth once for 6 days in the second cycle or the first cycle
  Interventions: Drug: Placebo; Dietary Supplement: fasting
- placebo tablets in postprandial (Active Comparator): placebo mimic iloperidone 1mg by mouth once for 6 days
  Interventions: Drug: Iloperidone 1 MG; Dietary Supplement: postprandial
- iloperidone in postprandial (Experimental): iloperidone 1mg by mouth once for 6 days
  Interventions: Drug: Placebo; Dietary Supplement: postprandial

INTERVENTIONS:
Drug: Iloperidone 1 MG — An open, random, two-period and two-sequence cross-test design was adopted for the fasting and postprandial groups, and the randomization method was adopted for each subject to randomly take the subjects or reference preparations.
  Arms: iloperidone in fasting; placebo tablets in postprandial
Drug: Placebo — An open, random, two-period and two-sequence cross-test design was adopted for the fasting and postprandial groups, and the randomization method was adopted for each subject to randomly take the subjects or reference preparations.
  Arms: iloperidone in postprandial; placebo tablets in fasting
Dietary Supplement: fasting — An open, random, two-period and two-sequence cross-test design was adopted for the fasting and postprandial groups, and the randomization method was adopted for each subject to randomly take the subjects or reference preparations.
  Arms: iloperidone in fasting; placebo tablets in fasting
Dietary Supplement: postprandial — An open, random, two-period and two-sequence cross-test design was adopted for the fasting and postprandial groups, and the randomization method was adopted for each subject to randomly take the subjects or reference preparations.
  Arms: iloperidone in postprandial; placebo tablets in postprandial

SUMMARY:
to inspect relevant pharmacokinetic parameters and relative exploitation degree, with fasting and postprandial dosing bioequivalence test under the condition of the human body, provide the basis for registration filing.

ELIGIBILITY:
Inclusion Criteria:

- 1) age above 18 years of age (including 18 years of age), male or female; 2) body mass index (BMI) = weight (kg)/height 2 (m2) , body mass index (including critical value) within 18~26 range; 3) health: no heart, liver, kidney, gastrointestinal tract, nervous system, mental disorder and metabolic abnormalities, such as history, physical examination showed the blood pressure, heart rate, ecg, respiratory system, liver, kidney, and normal or abnormal urinalysis performed without clinical significance; 4) subjects (including male subjects) are willing to take effective contraceptive measures in the next three months without pregnancy plan.

5) sign the informed consent before the test, and fully understand the contents, procedures and possible adverse reactions of the test; 6) be able to complete the research according to the test plan.

Exclusion Criteria:

- 1) HBsAg, HBeAg, HCV antibody, HIV antibody, and treponema pallidum are positive; 2) general physical examination, blood biochemistry, blood urine routine, serum prolactin and ECG examination are abnormal and have clinical significance; 3) past history or current in clinic with heart, breathing, endocrine, metabolism, kidney, liver, gastrointestinal tract, skin, infection, malignant tumor, blood and nerve system disease or mental/disorders; 4) take any medication, including over-the-counter and herbal medicines, within two weeks prior to the start of the trial; 5) the subjects' drinking history was more than 14 units of alcohol per week (1 unit = beer 285 mL, or liquor 25 mL, or wine 150 mL) or alcohol breath test was positive; 6) currently smoking >5 per day; 7) drug abuse or drug dependence or urine drug screening positive; 8) blood donation or a large amount of blood loss (>400 mL) or as a subject participating in drug trial sampling in the last three months; 9) underwent surgery within 4 weeks prior to the trial, or planned to perform surgical procedures during the study period; 10) test within 48 h before taking any special diet (including grapefruit, etc.), and/or contain xanthine diet or strenuous exercise, or other affect drug absorption, distribution, metabolism and excretion of food or drink, etc.; 11) drink excessive amounts of tea, coffee and/or caffeinated beverages (8 cups or more, 1 cup =250 mL) per day; 12) QTc period is greater than 450ms (male) or 470ms (female), or there is a history of QTc extension; 13) postural hypotension (the systolic blood pressure drops by 20mmHg or diastolic blood pressure drops by 10mmHg after standing on the supine position) 14) during the screening period or during the test, the female subjects were positive in lactation or pregnancy.

15) the researchers judged that the subjects' ability to comply with the research requirements was not necessarily complete or not necessarily able to comply with the subjects required by the test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-03-14 (Estimated)

PRIMARY OUTCOMES:
Cmax, | Change from Baseline afer dosing 0.33h,0.67h,1h,1.5h,2h,2.5h,3h,4h,6h,8h,12h ,24h,36h,48h,72h,96h,120h.
  Peak Plasma Concentration (Cmax) of iloperidone and metabolite P88
Tmax | Change from Baseline afer dosing 0.33h,0.67h,1h,1.5h,2h,2.5h,3h,4h,6h,8h,12h ,24h,36h,48h,72h,96h,120h.
  Tmax time to Peak Plasma Concentration (Cmax) of iloperidone and metabolite P88
AUC0-t、AUC0-∞ | Change from Baseline afer dosing 0.33h,0.67h,1h,1.5h,2h,2.5h,3h,4h,6h,8h,12h ,24h,36h,48h,72h,96h,120h.
  Area under the plasma concentration versus time curve (AUC) of iloperidone and metabolite P88
t1/2, | Change from Baseline afer dosing 0.33h,0.67h,1h,1.5h,2h,2.5h,3h,4h,6h,8h,12h ,24h,36h,48h,72h,96h,120h.
  t1/2, half-life period of iloperidone and metabolite P88
F | Change from Baseline afer dosing 0.33h,0.67h,1h,1.5h,2h,2.5h,3h,4h,6h,8h,12h ,24h,36h,48h,72h,96h,120h.
  F bioavalibility of iloperidone and metabolite P88
λz | Change from Baseline afer dosing 0.33h,0.67h,1h,1.5h,2h,2.5h,3h,4h,6h,8h,12h ,24h,36h,48h,72h,96h,120h.
  λz eliminating rate of iloperidone and metabolite P88

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of zhengzhou university., Zhengzhou, Henan, China